CLINICAL TRIAL: NCT06695728
Title: Hybrid Assistive Limb Effect on Jump Height: a Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Uskudar16
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Sport Injury
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid Assistive Limb Group (Experimental): exoskeleton
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — It consists of exercises to be done with the exoskeleton. These are; jumping exercise, squat, sit-stand and forward bending exercises.

SUMMARY:
The aim of this study is to investigate the effect of exercises performed with The Hybrid Assistive Limb device on the jump height of healthy non-athlete individuals.

DETAILED DESCRIPTION:
Cyberdyne Waist Type device will be worn by attaching 3 electrodes to the waist area and then attaching the device to the waist and legs with the help of belts. Then, the appropriate modes will be selected for the participant with the adjustments made on the device. It has 3 modes; CVC, the mode that produces torque value, that is, movement, according to muscle activation with only the bioelectric signals received from the person's skin. CAC, the mode that produces movement by presenting automatic values to the participant with data designed according to the specific software and algorithm of the device. CIC, the mode that produces movement completely according to the participant's control. In our study, investigators will produce movement according to the muscle activation created by the participant using the CVC mode. In this way, investigators will provide the brain-muscle relationship and motor learning parameters. The exercises will be applied for 30 minutes, 5 days a week, for a total of 40 sessions.

ELIGIBILITY:
Inclusion Criteria

* Being between 20 and 40 years old.
* Tall individuals over 120 cm (for accurate visual feedback in the assessment of jump height)
* Weighting less than 100 kg
* People who can perceive and follow the given instructions without any problems
* People who have not had any surgery in the last 6 months
* People who are not allergic to electrodes
* They should not have any skin tissue related disorders.
* People who do not use pacemakers
* People who do not have a history of seizures or a risk of seizures (epilepsy).
* They should not have heart and respiratory problems.
* People who have not experienced back pain in the last 3 months.
* People whose waist circumference is not more than 120 cm and whose thigh circumference is not more than 80 cm.
* No orthopedic or neurological problems that will affect the balance mechanism (e.g. Vertigo, cerebellum damage, ataxia).
* Not having used a Waist Type Hybrid Assistive Limb device before
* Not having worked with visual feedback devices such as Tecnobody D-Wall before
* Not having worked with any of the Cyberdyne Hybrid Assistive Limb devices before

Exclusion Criteria

* People with back pain or who have had surgery on their back
* Having had surgery within the last 6 months.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-02-23 (Actual)

PRIMARY OUTCOMES:
D-Wall (TecnoBody SRL, Italy) | 8 weeks
  D-Wall (TecnoBody SRL, Italy) is a digital mirror device consisting of a powerful platform paired with a control computer and a high-resolution 3D Kinect camera equipped with infrared beams that allow for motion capture. The system provides instant feedback on the patient's movements on a large LCD monitor, offering VR-based mirror therapy and game-based exercises.This device measures the jump height and the amount of power consumed. It records the data and presents the result numerically.

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Azizov, Study Chair — Uskudar University; Serhat Aslan, Study Chair — Uskudar University
Locations (1):
- Cybernıcx, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moll F, Kessel A, Bonetto A, Stresow J, Herten M, Dudda M, Adermann J. Use of Robot-Assisted Gait Training in Pediatric Patients with Cerebral Palsy in an Inpatient Setting-A Randomized Controlled Trial. Sensors (Basel). 2022 Dec 16;22(24):9946. doi: 10.3390/s22249946. PMID 36560316
- [Background] Watanabe H, Tsurushima H, Yanagi H. Effect of hybrid assistive limb treatment on maximal walking speed and six-minute walking distance during stroke rehabilitation: a pilot study. J Phys Ther Sci. 2021 Feb;33(2):168-174. doi: 10.1589/jpts.33.168. Epub 2021 Feb 13. PMID 33642694
- [Background] Matsuda M, Iwasaki N, Mataki Y, Mutsuzaki H, Yoshikawa K, Takahashi K, Enomoto K, Sano K, Kubota A, Nakayama T, Nakayama J, Ohguro H, Mizukami M, Tomita K. Robot-assisted training using Hybrid Assistive Limb(R) for cerebral palsy. Brain Dev. 2018 Sep;40(8):642-648. doi: 10.1016/j.braindev.2018.04.004. Epub 2018 Jul 14. PMID 29773349